CLINICAL TRIAL: NCT01182623
Title: Polyp Surface Pattern Recognition in the Identification of Neoplastic Polyps
Brief Title: The Value of Polyp Surface Pattern Recognition in the Identification of Neoplasia: a Prospective Study
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT2009/046
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Colonic Polyps
Keywords: FICE; Chromoendoscopy; Colonic polyps; Adenomas; Hyperplastic polyps
MeSH Terms: conditions — Colonic Polyps; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All polyps are sent for histological analysis as per standard protocol. This is not additional for the study and part of routine NHS practice. They will be kept and stored as per standard NHS protocols.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In vivo diagnosis: Patients undergoing colonoscopy where one or more polyps up to 10mm in size are found.
  Interventions: Other: Observation of surface patterns of polyps

INTERVENTIONS:
Other: Observation of surface patterns of polyps — examination of the surface patterns of polyps using FICE and indigo carmine dye spray

SUMMARY:
It is current practice to remove any polyps found during colonoscopy. This is because adenomatous polyps have the potential to turn into cancer. However, a proportion of polyps <10mm in size are hyperplastic, which cannot turn into cancer. Current practice requires these to be removed, as it is traditionally felt that they cannot be separated clinically from adenomas. This increases the risk of perforation and results in a significant cost in processing the samples. However, it has been suggested that it is possible to differentiate neoplastic from non neoplastic lesions using skills in polyp surface pattern recognition. If this is the case the investigators may be able to reduce the need for polypectomy The investigators believe that it is possible to tell the difference between polyps with cancerous potential and those that are harmless by assessment of surface patterns. This may enable us to improve the investigators clinical decisions when assessing polyps during colonoscopy, and reduce the number of unnecessary polypectomys being performed.

DETAILED DESCRIPTION:
Polyps are a common finding during colonoscopy. It is current practice to remove these lesions, as some have the potential to turn into cancer. However, not all polyps are the same. Polyps can be of three different types:

1. Hyperplastic, which have negligible potential to turn into cancer and if left would cause no harm. These account for around one third of all small polyps encountered
2. Adenomas, which can turn into cancer and should be removed
3. Polyp cancers, which should be either biopsied or removed completely

The management pathway for polyps >10mm is very simple as they are either likely to be adenomas which need removal or cancers which need a biopsy and tattoo. There is a rare possibility of these big polyps being hyperplastic / serrated adenomas and given the risk of malignant transformation, they need removal as well.

It has been traditionally felt that hyperplastic polyps cannot be separated clinically from adenomas or polyp cancers by the endoscopist. It is for this reason that all polyps are removed. However, polypectomy increases the risk of perforation and results in a significant cost in processing the samples. Recently it has been suggested that it is possible to differentiate neoplastic from non neoplastic lesions in the colon using skills in polyp surface pattern recognition.

Kudo's pit pattern is an effective way of in-vivo prediction of histology and differentiating neoplastic from non neoplasic polyps. However, it was originally described using vial staining which is cumbersome, time consuming and is not possible to perform outside Japan due to lack of availability and fears of toxicity related to gentian violet. It does however produce excellent results when used for pit pattern recognition. (Hurlstone DP C. S., 2004) It works by irreversibly binding microbial DNA and directly inhibiting cell replication. (Wakelin LPG, 1981).

Gentian violet is not the only way to examine the surface patterns of polyps. Many of the features can be seen with white light endoscopy. (Fu KI, 2004). Furthermore, there is extensive experience with other dies which are commonly used in Western Europe. Indigo carmine dye spray has been performed in studies in Japan, and has proven to be very effective in the assesment of polyp characteristics. It has been used for over 14 years in colonoscopy (Axelrad, 1996). Overall diagnostic accuracy by conventional view, chromoendoscopy and chromoendoscopy with magnification ranged from 68% to 83%, 82% to 92%, and 80% to 96%, respectively. (Axelrad AM, 1996) (Tung SY, 2001) (Eisen GM, 2002) (Su MY, 2004) (Apel D, 2006). It has the advantage over gentian violet that it does not bind to tissues and is therefore very safe. It has been questioned whether widespread applications of the techniques could influence the indications for biopsy sampling during colonoscopy and the indication for mucosectomy (Yasushi Sano, 2005).

When compared to standard colonoscopy, indigo carmine chromoendoscopy, with magnification, has been shown to increase the accuracy for polyp differentiation from 84% to 96% (Fu KI, 2004). High-resolution indigo carmine chromoendoscopy demonstrated a small increase in accuracy over chromoendoscopy without magnification from 81% to 83% . (Hurlstone DP K. M., 2005).

Because of its numerous benefits in lesion detection and assessment of polyps indigo carmine has become a standard part of colonoscopy and is recognised by the British Society of Gastroenterology as an important skill for the practicing endoscopist. It has become standard practice within Portsmouth Hospitals NHS trust when performing colonoscopy. This is a position which is reflected nationally in most large units which participate in the bowel cancer screening programme.

White light endoscopy and chromoendoscopy are not the only methods of examining colonic polyps. Computed virtual colonoscopy, where a video computer processor within the endoscopy equipment enhances the endoscopic picture have become commonly available. There are systems available from all of the main endoscope manufacturers, including narrow band imaging from Olympus and i-scan from Pentax. Fujinon has developed a very effective post processor technology called FICE which helps define the surface pattern of polyps in great detail. This is now a standard feature on all of the endoscopes produced by the company. It has been shown in a limited number of studies to offer a potentially useful alternative to dye spray in predicting in-vivo histology. (J. Pohl, 2008). A prospective randomised multicentre study looked at 764 patients with FICE compared to white light with targeted indigocarmine spray. It found that FICE and indigocarmine were both able to differentiate adenomas from neoplasia. There was a sensitivity in differentiating adenomas from non-neoplastic polyps of 92.7%,with FICE, comparable but not superior to that of indigocarmine (90.4%), with no statistically significant difference between the two techniques observed. (p=0.44.) FICE did not shorten the procedure time. A prospective series looking at FICE in the evaluation of colononic polyps up to 2cm in size by the same team suggested a sensitivity of 89% could be achieved. Unfortunately these studies looked at larger lesions and therefore it is difficult to say whether this could be achieved with polyps <1cm, where accurate assessment is clearly more difficult. However, it is in the smaller lesions where the greatest gain in terms of a change in management exists. (Pohl J N.-T. M., 2008).

It is generally accepted that further research is needed in this field. If it is possible for endoscopists to differentiate neoplastic from non neoplastic polyps the potential benefits both in terms of safety and histopathology costs would be significant. The current policy of polypectomy or biopsy of all polyps detected during colonoscopy is a very expensive option (£ 80-120) and carries a significant risk of perforation.

Within Portsmouth Hospitals NHS trust it has become standard practice to assess all polyps with FICE and dye spray with indigo carmine prior to removal. This is consistent with current guidelines from the British society of Gastroenterologists and is important both in the detection and assessment of polyps. These techniques are established and their importance in colonoscopy is not under investigation. What is unclear is whether endoscopists are able to differentiate neoplastic from non-neoplastic lesions on a basis of surface pattern recognition accurately enough to be able to change clinical practice.

We aim to assess the impact of surface pattern assessment on the potential management of patients, and whether it has the potential to safely replace the policy of biopsy / polypectomy for pateints with polyps <10mm in size.

ELIGIBILITY:
Inclusion Criteria:

* Patients found to have polyps up to 10 mm in size

Exclusion Criteria:

* Patient preference Clinicians judgement Obvious cancers Ulcerated polyps

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colonoscopy where one or more polyps are found.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2010-09-30 (Actual); Study Completion 2010-09-30 (Actual)

PRIMARY OUTCOMES:
The accuracy of predicted in-vivo polyp histology | 9 months

SECONDARY OUTCOMES:
• Sensitivity of white light endoscopy in predicting histology | 9 months
specificity of white light endoscopy in predicting histology | 9 months
Sensitivity of Chromoendoscopy in predicting histology | 9 months
Specificity of Chromoendoscopy in predicting histology | 9 months
Sensitivity of fujinon intelligent color enhancement (FICE) in predicting histology | 9 months
Specificity of fujinon intelligent color enhancement (FICE) in predicting histology | 9 months
Whether one technique is superior | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, MBBS,MD,MRCP, Principal Investigator — Consultant gastroenterologist
Locations (1):
- Portsmouth Hospitals NHS trust, Portsmouth, Hampshire, United Kingdom